CLINICAL TRIAL: NCT05108753
Title: Short-term Outcomes of Transanal Total Mesorectal Excision With Structured Training Curriculums in China: Retrospective Study of the First Twenty-five Cases in Seven High-volume Centers
Brief Title: Short-term Outcomes of Transanal Total Mesorectal Excision With Structured Training Curriculums in China
Status: Completed | Type: Observational
Sponsor: Shanghai Minimally Invasive Surgery Center (Other)
Responsible Party: Sponsor
Other Study IDs: MISC-TaTME-RETRO
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-11

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: 5 patients underwent TaTME under proctoring
  Interventions: Other: Procedure/Surgery
- Group 2: the first 10 patients underwent TaTME without proctoring
  Interventions: Other: Procedure/Surgery
- Group 3: the second 10 patients underwent TaTME without proctoring
  Interventions: Other: Procedure/Surgery

INTERVENTIONS:
Other: Procedure/Surgery — Transanal Total Mesorectal Excision

SUMMARY:
Transanal total mesorectal excision (TaTME) is an alternative for mid-low rectal cancer. In China, this procedure has been performed in high-volume centers with structured training curriculums. This study aimed to evaluate the short-term outcomes during the initial implementation of the TaTME procedure in high-volume centers who followed structured training curriculums in China.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years
* American Society of Anesthesiologists (ASA) score I to III
* A biopsy proven histological diagnosis of rectal carcinoma
* Undergoing transanal total mesorectal excision

Exclusion Criteria:

* Pregnant or lactating women
* Synchronous rectal carcinoma
* History of colorectal cancer or other malignant tumors
* Clinical evidence of metastasis
* Emergency procedure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: rectal cancer
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
incidence of anastomotic leakage | thirty days after surgery
  according to the International Rectal Cancer Study Group

SECONDARY OUTCOMES:
incidence of Defecation disorders | 6 months after surgery
  A Wexner score >10 indicated the existence of defecation dysfunction
incidence of positive distal resection margin | 30 days after surgery
  A positive distal resection margin (DRM) was diagnosed with the presence of tumor cells within 1mm from the DRM
incidence of positivecircumferential resection margin | 30 days after surgery
  The positive circumferential resection margin (CRM) was defined as the presence of tumor cells within 1 mm from the CRM

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Ruijin Hospital, Shanghai, Shanghai Municipality
  - Shanghai Minimally Invasive Surgery Center, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided